CLINICAL TRIAL: NCT05834569
Title: The Impact of Intravenous Administration of Perioperative Acetaminophen and Ibuprofen Combination (Maxigesic®) on Postoperative Delirium in Elderly Patients Undergoing Minimally Invasive Lung Segmentectomy or Lobectomy
Brief Title: Impact of Maxigesic on Delirium After Minimally Invasive Lung Surgery in Elderly Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated early owing to challenges in completing the research registration process.
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Kyongbo Pharmaceutical Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, Kim, Heezoo, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023GR0023
Record Dates: First submitted 2023-03-07; First posted 2023-04-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Delirium; Aged; Lung Neoplasms; Robotic Surgical Procedures; Thoracic Surgery, Video-Assisted
Keywords: Postoperative delirium; Elderly; Minimally invasive surgery; Lung segmentectomy; Lung lobectomy
MeSH Terms: conditions — Delirium; Lung Neoplasms; Emergence Delirium | interventions — Acetaminophen; Ibuprofen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maxigesic group (Experimental)
  Interventions: Drug: Acetaminophen and Ibuprofen
- Control group (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Acetaminophen and Ibuprofen — Patients in the Maxigesic group will be administered a total of 5 doses of the drug (20mg/kg, maximum dose per serving: 1g) every 6 h from immediately after anesthetic induction.
  Arms: Maxigesic group
Drug: Normal saline — Patients in the control group will be administered equal amounts of normal saline at the same time points.
  Arms: Control group

SUMMARY:
The primary aim of this interventional study is to investigate the impact of perioperative administration of Maxigesic (combination of acetaminophen and ibuprofen) on delirium after minimally invasive lung surgery in elderly patients. The Maxigesic group receives a total of 5 doses of Maxigesic (20mg/kg, maximum dose per serving: 1g) every 6 h from immediately after anesthesia induction. The control group receives the same volume of normal saline. Researchers compare the incidence and severity of postoperative delirium for 5 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older undergoing minimally invasive lung lobectomy or segmentectomy

Exclusion Criteria:

* Hypersensitivity to the main ingredients and additives of Maxigesic
* Hypersensitivity to aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs)
* Alcoholism / Alcohol intoxication
* Severe hematological abnormalities
* Bleeding tendency (e.g., Spontaneous bleeding)
* Severe hepatic dysfunction (AST, AST ≥2.5 * upper normal limit(UNL) or Total bilirubin ≥3.0 mg/dl)
* Severe renal dysfunction (eGFR <30 ml/min/1.73m2 or Dialysis)
* Severe heart failure (Left ventricle ejection fraction <30%)
* Uncontrolled hypertension(HTN) (Systolic blood pressure >180 mmHg)
* Symptomatic asthma in need of treatment
* Anticoagulants or antiplatelet agents are maintained for up to 5 days before surgery
* Barbiturates or tricyclic antidepressants (TCAs)
* High-dose methotrexate (MTX) for cancer treatment
* Preoperative cognitive impairment, dementia, or delirium
* Inability to understand the research and instructions for this study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium(POD) | From immediately after surgery to 5 days after surgery
  Confusion assessment method(CAM)/Confusion Assessment Method for the ICU (CAM-ICU) or delirium record on electrical medical record(EMR) will be used for the evaluation of POD.

SECONDARY OUTCOMES:
Severity of POD | From immediately after surgery to 5 days after surgery
  CAM-S(severity) will be utilized to assess the severity of POD. (*CAM-S is measured on 0-7 (short form) and 0-19 (long form) scale, and the higher the score, the greater the POD severity.)
Duration of POD | From immediately after surgery to 5 days after surgery
  CAM/CAM-ICU or delirium record on EMR will be used to estimate the duration of POD.
Preoperative cognition | 1 day before surgery
  Mini-mental state examination(MMSE) will be used to evaluate the participants' preoperative cognition. (*MMSE is measured on 0-30 scale, and the lower the score, the more cognitively impaired the patient is.)
Preoperative cognition | 1 day before surgery
  Montreal cognitive assessment(MoCA) will be used to evaluate the participants' preoperative cognition. (*MoCA is measured on 0-30 scale, and the lower the score, the more cognitively impaired the patient is.)
Preoperative frailty | 1 day before surgery
  Clinical frailty scale(CFS) will be utilized to assess the preoperative frailty (*CFS is used to determine comprehensive geriatric assessment. It is measured on 1-9 scale, and the higher the scale, the more frail the patient is.)
Postoperative pain | Immediately after surgery to postoperative 48 hours
  Numerical rating scale (NRS) or Visual analogue scale (VAS) will be used to determine the postoperative pain severity (*NRS and VAS are measured on a 0-10 scale, and the higher the score, the more severe the patient's pain. If the patient can verbalize their pain, use the NRS; otherwise, use the VAS to assess pain).
Consumption of opioids | Immediately after surgery to postoperative 48 hours
  Opioid consumption is measured by converting them into morphine equivalents.
Postoperative nausea, vomiting | Immediately after surgery to postoperative 48 hours
  Nausea is measured by scoring on a scale of 0-10. The higher the score, the more severe the symptom. Whether the patients vomit or not is observed and recorded.
ICU stay | Immediately after surgery to ICU discharge(usually within about 5 days after surgery)
  Determine how many days the participant stays in the ICU.
Hospital stay | Immediately after surgery to hospital discharge(usually within about 30 days after surgery)
  Determine how many days the participant stays in the hospital.
Postoperative complications | Immediately after surgery to hospital discharge(usually within about 30 days after surgery)
  Investigate all kinds of complications that occur after surgery.
Drug side effects | Immediately after surgery to hospital discharge(usually within about 30 days after surgery)
  Investigate complications suspected to be side effects caused by the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Heezoo Kim, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The investigators have no plans yet to share individual participant data (IPD) with other researchers.